CLINICAL TRIAL: NCT03124017
Title: Electronic Alert System Combined With a Risk Score Calculation Tool for Improving Appropriate Thromboprophylaxis in Hospitalized Medical Patients: a Randomized Controlled Trial
Brief Title: Electronic Alert System for Improving Thromboprophylaxis in Hospitalized Medical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 159/14
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Alert Group (Experimental): Electronic alert and the Geneva Risk Score calculation tool issued in the electronic patient chart
  Interventions: Other: Electronic alert and the Geneva Risk Score calculation tool issued in the electronic patient chart
- Control Group (No Intervention): No electronic alert and no Geneva Risk Score calculation tool issued in the electronic patient chart

INTERVENTIONS:
Other: Electronic alert and the Geneva Risk Score calculation tool issued in the electronic patient chart
  Arms: Alert Group

SUMMARY:
The investigators aim to investigate whether a computer-based alert system in the electronic patient chart and order entry system using the Geneva Risk Score as clinical decision support tool to estimate the risk of venous thromboembolism improves the rate of appropriate thromboprophylaxis among hospitalized medical patients.

DETAILED DESCRIPTION:
The use of thromboprophylaxis among acutely ill hospitalized medical patients remains inconsistent. The present study aims to improve the use of appropriate thromboprophylaxis by implementing a computer-based alert system combined with a Geneva Risk Score calculation tool in the electronic patient chart and order entry system. Consecutive acutely ill medical patients without indication for therapeutic anticoagulation or ongoing therapeutic anticoagulant treatment admitted to the medical wards of the University Hospital Bern, Switzerland, will be randomized in a 1:1 fashion to the alert group in which an alert and the Geneva Risk Score calculation tool will be issued in the electronic patient chart or to the control group in which no alert will be issued. The primary endpoint is the rate of appropriate thromboprophylaxis during hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Acutely ill medical patients admitted to medical wards

Exclusion Criteria:

* Indication for therapeutic anticoagulation or ongoing therapeutic anticoagulant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1756 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Rate of appropriate thromboprophylaxis | During hospital stay (expected average duration of 1 week)

SECONDARY OUTCOMES:
Use of the Geneva Risk Score calculation tool by the physician in charge | During hospital stay (expected average duration of 1 week)
Rate of correct calculation of the Geneva Risk Score through the calculation tool by the physician in charge | During hospital stay (expected average duration of 1 week)

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kucher, Prof. M.D., Principal Investigator — Swiss Cardiovascular Center, Division of Vascular Medicine, University of Bern, University Hospital Bern, Bern, Switzerland
Locations (1):
- Swiss Cardiovascular Center, Inselspital, University of Bern, Bern, Switzerland

REFERENCES:
- [Derived] Spirk D, Stuck AK, Hager A, Engelberger RP, Aujesky D, Kucher N. Electronic alert system for improving appropriate thromboprophylaxis in hospitalized medical patients: a randomized controlled trial. J Thromb Haemost. 2017 Nov;15(11):2138-2146. doi: 10.1111/jth.13812. Epub 2017 Sep 20. PMID 28836340